CLINICAL TRIAL: NCT05284630
Title: Evaluation of the Effect of Exercise Program Followed by Mobile Application on Pain, Quality of Life, Functionality and Stability in the Treatment of Patients With Chronic Neck Pain
Brief Title: Using Mobile Application for Rehabilitation in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Medical Park Hospital Istanbul (Other)
Responsible Party: Principal Investigator, Mehmet Burak Uyaroğlu, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaglikBilimU
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neck Pain; Chronic Pain
Keywords: Neck Pain; Chronic Pain; mobile Health; Mobile Apps; Quality of Life
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Exercise; Electric Stimulation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): Exercise follow up with mobile application in patients with chronic neck pain five sessions a week for 4 weeks
  Interventions: Other: Exercise follow up with mobile application; Procedure: Electrotherapy
- Control Group (Active Comparator): Home based exercise follow up him/herself in patients with chronic neck pain five sessions a week for 4 weeks
  Interventions: Other: Home-Based Exercise Program followed by paper booklet; Procedure: Electrotherapy

INTERVENTIONS:
Other: Exercise follow up with mobile application — Exercises will be followed by mobile application. Electrotherapy will be performed.
  Other Names: Exercise with Mobile Application
  Arms: Experimental Group
Other: Home-Based Exercise Program followed by paper booklet — Exercise will be followed by paper booklet. Electrotherapy will be performed.
  Arms: Control Group
Procedure: Electrotherapy — Electrotherapy will be performed.

SUMMARY:
The aim of this study is to reduce pain, increase range of motion, increase the endurance of deep cervical flexors muscles, and increase quality of life with mobile application in the treatment of patients with chronic neck pain. Although many benefits of exercises have been proven, the effectiveness, follow-up and continuity of exercise will be investigated with mobile application tracking.

DETAILED DESCRIPTION:
One of the important factors in mechanical chronic neck pain is the decrease in the endurance of the deep cervical flexor muscles. As a result of this decrease, an increase to the activation of M. Scalenus Anterior and M. Sternocleidomastoid muscles is observed. It is known that patients avoid some movements due to pain, and as a result, loss of muscle strength and endurance in the neck, upper back, around the scapula and shoulder occurs. The loss in strength and endurance, combined with the severity of pain, may affect the stability of the upper extremity has been considered.

Patients with chronic neck pain may experience a number of problems due to the predisposition to accompany pain or some problems caused by neck pain. It is known that all these problems affect the quality of life of patients by limiting their daily living activities.

With the developing technology, mobile health applications have started to be used more and more in our lives. In addition to preventing disease, reducing risk factors, increasing physical activity and quality of life, mobile applications are used in many different areas such as diagnosis, treatment, feedback and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic neck pain in the past 6 months
* No communication problem
* Be Literate,
* Individuals who speaks Turkish and can use developed mobile application

Exclusion Criteria:

* Previous neck or shoulder surgery,
* Shoulder pain due to any reason,
* Having tumor or inflammatory disease underlying neck pain
* Having mental disorder,
* Individual with sequestered disc level or root compression,
* Individual with uncontrolled diabetes mellitus and hypertension
* Patients received additional treatment
* Patients who did not complete physical therapy sessions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Change from pre-interventional Neck Disability Index score at the end of the intervention that will be performed 5 days in a week at a total of 4 weeks.
  The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation.

SECONDARY OUTCOMES:
Visual Analog Scale | Change from pre-interventional Visual Analog Scale score at the end of the intervention that will be performed 5 days in a week at a total of 4 weeks.
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain).
Assessment of the degree of joint range of motion | Change from pre-interventional Range of Motion Assesment score at the end of the intervention that will be performed 5 days in a week at a total of 4 weeks.
  Active range-of-motion(ROM)as measured by a goniometer A ROM assessment is most commonly used to measure movement of the ankles, knees, hips, shoulders, elbows, wrists and fingers. Measures are taken on consecutive occasions to assess any change over time. They are used to determine whether an individual's ROM is within the expected range.
Manual Muscle Test | Change from pre-interventional Manual Muscle Test Assesment score at the end of the intervention that will be performed 5 days in a week at a total of 4 weeks.
  An assessment of muscle strength is typically performed as part of a patient's objective assessment and is an important component of the physical exam.
  This test involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly.
The System Usability Scale (SUS) | Change from pre-interventional System Usability Scale score at the end of the intervention that will be performed 5 days in a week at a total of 4 weeks.
  The System Usability Scale (SUS) provides a "quick and dirty", reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Originally created by John Brooke in 1986, it allows you to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Akçay, PT,MSc, Study Chair — Saglik Bilimleri Universitesi; Gamze Koyutürk, PT,MSc, Principal Investigator — Saglik Bilimleri Universitesi; Mehmet Burak Uyaroğlu, PT,MSc, Study Chair — Saglik Bilimleri Universitesi; Dudu Kübra Akyol, PT, Study Chair — IAU Medical Park Florya Hospital; Emre Serdar Atalay, Ass. Prof., Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Saglık Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No